CLINICAL TRIAL: NCT06103084
Title: Acceptability and Effectiveness of Local Food Solutions for the Prevention of Acute Malnutrition in Tigray, Northern Ethiopia (ELOFSAM)
Brief Title: Effectiveness of Local Food Solutions for the Prevention of Acute Malnutrition in Tigray, Northern Ethiopia (ELOFSAM)
Acronym: ELOFSAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mekelle University (Other)
Collaborators: Tigray Development Association (Unknown); Mums for Mums (Unknown); Tigray Health Research Institute (Unknown); Tigray Health Bureau (Unknown); UNICEF Tigray Office (Unknown)
Responsible Party: Principal Investigator, Afework Mulugeta, Professor, Mekelle University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MUCHS
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acute Malnutrition in Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bahgina group (Experimental): The Bahgina treatment group will be supplemented with Bahgina, a locally produced cereal based product for a maximum of six months at 200g/day.
  Interventions: Dietary Supplement: Bahgina
- SQLNS group (Experimental): The small quantity lipid based nutrient supplements (SQLNS) group will be provided with 20g of SQLNS/day for a maximum of six months.
  Interventions: Dietary Supplement: SQLNS
- Control (No Intervention): The control group will get nothing except the routine nutrition services and products provided by the local government sectors.

INTERVENTIONS:
Dietary Supplement: Bahgina — Bahgina, a locally produced cereal based food, will be provided at 200g/day/child for a duration of six months on top of the routine nutrition services provided by the local government and nutrition partners.
  Arms: Bahgina group
Dietary Supplement: SQLNS — Small quantity lipid based nutrient supplement (SQ-LNS) will be provided at 20g/day/child for a duration of six months on top of the routine nutrition services provided by the local government and nutrition partners.
  Arms: SQLNS group

SUMMARY:
The lack of diversified and enriched complementary foods is one of the key causes of the high burden of acute malnutrition among 6-23 months old children in Ethiopia. Thus, a new innovative way of diversifying and enriching complementary foods is essential in communities where vulnerable populations are likely to have nutrient gaps in their typical diets and multiple micronutrient deficiencies. The purpose of this project is to investigate the acceptability and effectiveness of locally produced cereal based foods (LP-CBFs) and small quantity lipid based nutrient supplements (SQ-LNS) as preventive interventions to effectively reduce the burden of acute malnutrition among 6-23 months old children in the post conflict settings of Tigray, Northern Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* All 6-23 months old children

Exclusion Criteria:

* 6-23 months old children with severe acute malnutrition.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7530 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Acute Malnutrition | six months
  The burden or prevalence of acute malnutrition among 6-23 months old children.

CONTACTS AND LOCATIONS:
Overall Officials: Hayelom Kahsay, MD, Study Chair — Tigray Health Research Institute
Locations (1):
- Tigray Health Research Institute, Mek'ele, Tigray, Ethiopia